CLINICAL TRIAL: NCT03418740
Title: Neurological Measures of Progression in Children With Friedrich Ataxia
Brief Title: Neurology Measures in FA Children
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Florida (Other); University of California, Los Angeles (Other); Food and Drug Administration (FDA) (U.S. Federal Agency); Friedreich's Ataxia Research Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: 17-014390; FD006029-01 (Other Grant/Funding Number: FDA)
Record Dates: First submitted 2018-01-26; First posted 2018-02-01 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Friedreich Ataxia
Keywords: Friedreich; Ataxia; FRDA; FA; Friedrich Ataxia (FRDA)
MeSH Terms: conditions — Friedreich Ataxia; Ataxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Whole blood and plasma to measure frataxin protein and other present biomarkers.
  Buccal cells (inner cheek cells) to measure frataxin protein levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FA Children: Children between the ages of 2 and 18 with genetically confirmed Friedreich's Ataxia

SUMMARY:
The purpose of this study is to identify ways to follow progression of Friedreich's Ataxia (FA) and be able to measure changes over time in children with FA. Participants will have biannual visits to observe how the disease progresses over time and determine the rate of progression.

Funding Source- Food and Drug Administration Office of Orphan Products Development (FDA OOPD).

DETAILED DESCRIPTION:
Investigators seek to identify biological and clinical tests to be used in future clinical trials. The purpose of this research study is to learn more about Friedreich's Ataxia (FA) progression in children. There will be biannual visits which will include a core set of tests and procedures. These include: a collection of medical history, detailed neurological exam, ataxia scales, and health questionnaires. At each visit, blood and cheek swab samples will be obtained to monitor frataxin levels.

A select number of Children's Hospital of Philadelphia (CHOP) participants will have the opportunity to participate in further procedures to better understand how FA affects different tissues. These include a Magnetic Resonance Imaging (MRI) scan and a Motor Evoked Potentials (MEP) procedure.

The MRI scan analyzes how muscle activity is affected in FA. The magnet will be used to capture images of the calf muscle before and after exercising on an ergonomic foot pedal.

The MEP procedure measures how strong the connection is between the brain's motor cortex and a selected body part, specifically the participant's dominant hand.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 2 to 18 years.
2. Genetically confirmed diagnosis of Friedreich's Ataxia (FA) or clinically confirmed diagnosis of FA, pending confirmatory genetic testing through a commercial or research laboratory
3. Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria:

1) Inability to complete study evaluations

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will primarily take place at the Children's Hospital of Philadelphia (CHOP), with a select number of subjects only participating in the clinical testing at the University of Florida and University of California Los Angeles (UCLA). The investigators expect to recruit approximately 100 children across all three sites and study each of them over a 3 year period. Children with a genetically or clinically confirmed diagnosis of Friedreich's Ataxia (FA) will be offered participation.
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Lynch, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (3):
- United States (3):
  - University of California, Los Angeles, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall, among 108 individuals enrolled, 19 were excluded from the analysis population for one or more reasons. These included missing mFARS data at baseline or follow-up, early disease stage, and inability to ambulate at baseline.
Groups:
- FA Children: The present study enrolled 108 children aged 6.7 to 18y with genetically confirmed FRDA (Friedreich Ataxia) between Oct 2017 and October 2019.
Period: Overall Study
Arm/Group | FA Children
Started | 108
Number of Participants in the Analysis Population | 89 (Despite description that completed population was 85, the number 89 more accurately captures the analysis group since some subjects were excluded for multiple reasons.)
Completed | 85
Not Completed | 23
Not completed — Lost to Follow-up | 13
Not completed — Scheduling Issues | 7
Not completed — Withdrawal by Subject | 2
Not completed — Unable to Continue Consent | 1

BASELINE CHARACTERISTICS:
Population: Overall, among 108 individuals enrolled, 19 were excluded from the analysis population for one or more reasons.
Groups:
- FACHILD: The population enrolled in this study was a young, severely affected cohort, indicated by high GAA1 repeat lengths and early ages of onset. It was a mixed early/typical FRDA population, suggesting a certain level of diversity despite tight pediatric enrollment criteria.
Arm/Group | FACHILD
Number analyzed (Participants) | 89
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.3 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 41
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 89
mFARS Total (93) [Mean (Standard Deviation); unit: units on a scale] — The modified Friedreich's Ataxia Rating Scale (mFARS) is a clinically validated set of assessments that measures disease progression in neurological disorder Friedreich Ataxia. The mFARS consists of four sections: bulbar (FARS A), upper limb coordination (FARS B), lower limb coordination (FARS C), and upright stability (FARS E). Minimum score of 0 in each section represents minimal disease affect. Maximum scores vary per section, with higher scores corresponding to more severe disease affect in that section. Maximum composite mFARS score 93 derived from total combined subsection scores.
  units on a scale | 37.8 (11.7)
Upright Stability (FARS E, 36) [Mean (Standard Deviation); unit: units on a scale] — Subsection E in the mFARS assesses upright stability as a neurologic component of Friedreich Ataxia. Minimum score of 0 represents minimal effect in upright stability. Maximum score of 36 denotes severe effect and loss of coordination to perform exam tasks.
  units on a scale | 22.3 (5.3)
Upper Limbs (FARS B, 36) [Mean (Standard Deviation); unit: units on a scale] — Subsection B in the mFARS assesses upper limb function as a neurologic component of Friedreich Ataxia. Minimum score of 0 represents minimal effect in upper limb coordination. Maximum score of 36 denotes severe effect and no coordination to perform exam tasks.
  units on a scale | 9.2 (5.3)
Lower Limbs (FARS C, 16) [Mean (Standard Deviation); unit: units on a scale] — Subsection C in the mFARS assesses lower limb function as a neurologic component of Friedreich Ataxia. Minimum score of 0 represents minimal effect in lower limb coordination. Maximum score of 16 denotes severe effect and no coordination to perform exam tasks.
  units on a scale | 5.9 (2.4)
Bulbar Function (FARS A, 5) [Mean (Standard Deviation); unit: units on a scale] — Subsection A in the mFARS assesses bulbar function as a neurologic component of Friedreich Ataxia. Minimum score of 0 represents minimal affect in speech or cough. Maximum score of 5 denotes severe affect and almost no useful speech and nearly absent or total loss of ability to cough.
  units on a scale | 0.3 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in mFARS (Modified Friedreich's Ataxia Rating Scale) Score
Description: The Friedreich Ataxia Rating Scale (FARS) measures neurological function in FA. It is a composite measure reflecting neural substrates with five-subscales (sections A to E), measuring bulbar function, upper limb coordination, lower limb coordination, peripheral nerves, and upright stability. The modified FARS (mFARS) shortens the bulbar subscale to 2 items and excludes the peripheral nerve subscale.
  Total scoring is a summation of subscales, with a maximum score of 93 points for mFARS and 125 for FARS. The mFARS score ranges for each subscale are: Bulbar: 0 - 5, Upper Limb: 0 - 36, Lower Limb: 0 - 16, Upright Stability: 0 - 36.
  The overall change in mFARS and its sub scores across 3 years was the outcome measure analyzed at 0, 1, 2, and 3 year visits. Each subsection has a minimum score of 0, indicating minimal effect for that component. Maximum values per section vary based on the tasks performed in each subsection; a higher score indicates greater dysfunction on that component.
Time Frame: Baseline up to 36 Months
Population: Among 108 individuals enrolled,19 were excluded from the analysis population for one or more concurrent reasons. These included missing mFARS data (baseline or follow-up, n = 6), early disease stage (n = 3, mFARS baseline values 1, 7, 12.3), and inability to ambulate at baseline (n = 13).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- FA Children: Children between the ages of 6 and 18 with genetically confirmed Friedreich's Ataxia
Arm/Group | FA Children
Number analyzed (Participants) | 89
units on a scale
  mFARS 1Y | 2.9 [1.6 to 4.2]
  mFARS 2Y | 4.9 [3.6 to 6.3]
  mFARS 3Y | 7.7 [6.4 to 9.0]
  FARS E 1Y | 2.2 [1.5 to 2.9]
  FARS E 2Y | 3.7 [3.0 to 4.5]
  FARS E 3Y | 5.5 [4.7 to 6.2]
  FARS B 1Y | 0.3 [-0.4 to 1.1]
  FARS B 2Y | 0.3 [-0.4 to 1.1]
  FARS B 3Y | 0.6 [-0.1 to 1.3]

2. Secondary Outcome: Change in Timed 25-Foot Walk (T25FW) Test
Description: The timed 25-foot walk (T25FW) test examines gait speed. The participant walks the distance of 25 feet as fast and safe as possible. Participants may use assistive devices during this task. The T25FW test was analyzed at 0, 1, 2, and 3 year visits.
Time Frame: Baseline up to 36 Months
Population: Walking tests were carried out in the order: T25FW (twice), 1MW (twice), 6MW, and TUG. The T25FW, was most consistently performed at Baseline. Number of participants analyzed decreased after baseline at year 1, 2, and 3 as subjects were unable to complete the test. Reasons for not performing a test were missed visits, and, if assessment was performed, devices used.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | FA Children
Number analyzed (Participants) | 51
seconds
  T25FW 1Y | -0.2 [-0.3 to -0.1]
  T25FW 2Y: number analyzed (Participants) | 37
  T25FW 2Y | -0.4 [-0.5 to -0.3]
  T25FW 3Y: number analyzed (Participants) | 35
  T25FW 3Y | -0.5 [-0.6 to -0.4]

3. Secondary Outcome: Change in 9-Hole Peg Test (9HPT)
Description: This test examines finger dexterity and involves placing and removing nine pegs in a pegboard and then removing them in the quickest possible time. The 9HPT has high intra- and inter-rater reliability and is the most commonly used measure of upper limb function in FA. The 9HPT was analyzed at 0, 1, 2, and 3 year visits.
Time Frame: Baseline up to 36 Months
Population: The number of participants analyzed decreased after baseline at years 1, 2, and 3 as subjects were unable to complete the test. Reasons for not performing a test were missed visits or refusal to complete task.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | FA Children
Number analyzed (Participants) | 61
seconds
  9HPT 1Y | -0.1 [-0.2 to -0.1]
  9HPT 2Y: number analyzed (Participants) | 47
  9HPT 2Y | -0.2 [-0.3 to -0.2]
  9HPT 3Y: number analyzed (Participants) | 54
  9HPT 3Y | -0.3 [-0.3 to -0.2]

4. Secondary Outcome: Change in Timed Up and Go (TUG) Test
Description: The Timed Up and Go (TUG) test is a timed measure during which the participant has to stand up from a chair, walk 3 meters, turn around, walk back, and sit down. The participant is asked to perform the task as fast and as safe as possible. The TUG is a norm-referenced measure that has established reliability for quickly assessing functional ambulatory mobility and dynamic balance in adults and children. The TUG test was analyzed at 0, 1, 2, and 3 year visits.
Time Frame: Baseline up to 36 Months
Population: The TUG was assessed last and was performed by a higher proportion of patients vs. the 6MW. As the difficulty of the tests increased the amount of missing data increased, consistent with the progressive nature of FRDA. The number of participants analyzed decreased after baseline at years 1, 2, and 3 as subjects were unable to complete the test. Possible reasons for not performing a test were collected as "fatigue", "refused", "unable" and "unable, unrelated to disease progression".
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | FA Children
Number analyzed (Participants) | 28
seconds
  TUG*100 1Y | -1.4 [-2.3 to -0.5]
  TUG*100 2Y: number analyzed (Participants) | 22
  TUG*100 2Y | -3.6 [-4.6 to -2.6]
  TUG*100 3Y: number analyzed (Participants) | 22
  TUG*100 3Y | -4.9 [-5.9 to -3.9]

5. Secondary Outcome: Change in Berg Balance Scale (Full Length) (BBS) Score
Description: The Berg Balance Scale (BBS) is a widely used assessment to determine a person's balance abilities. The BBS includes a 14-item scale with static and dynamic activities of varying difficulty. The overall change in BBS score across 3 years was analyzed at 0, 1, 2, and 3 year visits. Scoring is based on a summation of the 14 item tasks scored on a five-point scale, with a range of 0-4 for each task.
  0 = lowest level of function 4 = highest level of function. Highest possible score = 56 A score of < 45 indicates a greater risk of falling.
Time Frame: Baseline up to 36 Months
Population: The number of participants analyzed decreased after baseline at years 1 and 2 as subjects were unable to complete the test. Reasons for not performing a test were missed visits, and refusal to complete task.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | FA Children
Number analyzed (Participants) | 49
units on a scale
  BBS 1Y: number analyzed (Participants) | 44
  BBS 1Y | -6.5 [-9.1 to -3.9]
  BBS 2Y: number analyzed (Participants) | 42
  BBS 2Y | -10.4 [-13.0 to -7.7]
  BBS 3Y | -15 [-17.6 to -12.5]

6. Secondary Outcome: Change in FA-Activities of Daily Living Scale (ADL) Score
Description: The Activities of Daily Living (ADL) assesses functional status as a measurement of the participant's ability to perform activities of daily living independently. The ADL comprises 9 questions, each question scored on a scale of 0 to 4, though participants may use increments of 0.5 if they feel they fall between two items. As with the mFARS, the total ADL score is comprised of a summation of each scored question. A minimum value of 0 on the ADL scale indicates self-evaluation of minimal effect for neurological disease components. A maximum score of 36 on the ADL indicates most severe self-evaluation of symptoms included on the survey. The overall change in ADL score across 3 years was analyzed at 0, 1, 2, and 3 year visits.
Time Frame: Baseline up to 36 Months
Population: The number of participants analyzed decreased after baseline at years 1, 2, and 3 as subjects were unable to complete the test. Reasons for not performing a test were missed visits, and refusal to complete task.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | FA Children
Number analyzed (Participants) | 70
units on a scale
  ADL 1Y | 0.1 [-0.7 to 0.9]
  ADL 2Y | 1.9 [1.1 to 2.7]
  ADL 3Y: number analyzed (Participants) | 66
  ADL 3Y | 3 [2.2 to 3.9]

7. Secondary Outcome: Change in 1-minute Walk (1MW) and 6-minute Walk (6MW) Tests
Description: The Timed 1-minute Walk (T1MW) and timed 6-minute Walk are quantitative mobility and leg function performance tests based on distance traveled in one minute and six minutes. The participant is directed to one end of a clearly marked course and is instructed to walk back and forth as quickly as possible for one minute. The task is then repeated for six minutes. The distance is calculated by measuring how far the participant travels along the marked course.
Time Frame: Baseline up to 36 Months
Population: Walking tests were carried out in the order: T25FW (twice), 1MW (twice), 6MW, and TUG. There was a notable increase in fatigue and refusals to complete the longer walking tests after the first trial of the 1MW, followed by the 6MW. As the difficulty of the tests increased the amount of missing data increased, consistent with the progressive nature of FRDA. Possible reasons for not performing a test were collected as "fatigue", "refused", "unable" and "unable, unrelated to disease progression".
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | FA Children
Number analyzed (Participants) | 33
meters
  1MW 1Y | -11 [-15.7 to -6.2]
  1MW 2Y: number analyzed (Participants) | 28
  1MW 2Y | -15.7 [-20.8 to -10.7]
  1MW 3Y: number analyzed (Participants) | 30
  1MW 3Y | -23.1 [-28.0 to -18.1]
  6MW 1Y: number analyzed (Participants) | 20
  6MW 1Y | -13.1 [-56.0 to 29.7]
  6MW 2Y: number analyzed (Participants) | 11
  6MW 2Y | -65.8 [-120.3 to -11.4]
  6MW 3Y: number analyzed (Participants) | 8
  6MW 3Y | -67.4 [-129.9 to -4.9]

ADVERSE EVENTS:
Time Frame: Adverse events were not collected as part of this study. All-Cause Mortality was assessed through study completion, up to 2 years.
Description: Adverse events were not collected as part of this study. There was one subject death on the study that was attributed to complications of their disease.
Groups:
- FA Children: The present study enrolled 108 children aged 6.7 to 18y with genetically confirmed FRDA between Oct 2017 and October 2019. Twenty-three individuals withdrew from the study before the final visit. Of those, 13 were lost to follow-up, 7 were unwilling/unable to commit enough time (due to the tight visit schedule), 2 withdrew for other reasons (related to the pandemic/travelling), and 1 was unable to continue consent.
  Adverse events were not collected on this study.
Arm/Group | FA Children
All-Cause Mortality (participants affected / at risk) | 1/89
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Potential training effects of the repeated outcome measures as well as placebo effects might have increased variability. Varying demographic and genetic factors such as the presence of point mutations, GAA1 repeat length, age of onset and age at baseline also contribute to variability and may impact the rates of change over time. The COVID-19 epidemic also contributed to intermittent loss of data, and supplementing with virtual visits had limited value.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/40/NCT03418740/Prot_SAP_000.pdf